CLINICAL TRIAL: NCT03442920
Title: The Effects of Obesity and Periodontitis on Biochemical Parameters in Women Subjects
Brief Title: Evaluation of Periodontal Diseases and Obesity in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Esra Guzeldemir-Akcakanat, Professor, Kocaeli University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 114S144
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Periodontal Diseases; Obesity
Keywords: obesity; periodontal diseases; gingival crevicular fluid; saliva; serum
MeSH Terms: conditions — Periodontal Diseases; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese women (Experimental): Obese women who participated exercise programme.
  Interventions: Other: Exercise
- Normal weighted (No Intervention): Normal weighted women with non-periodontitis

INTERVENTIONS:
Other: Exercise — This group made exercise for 12 week/3 times a week.
  Arms: Obese women

SUMMARY:
The aim of this study was to evaluate the effect of obesity and exercise on periodontal and biochemical parameters [serum, saliva and gingival crevicular fluid (GCF) adipokines (interleukin-1β, tumor necrosis factor-α, leptin, resistin and adiponectin)].

DETAILED DESCRIPTION:
It is thought that adipokines may play a role on periodontal disease in obese subjects, periodontal disease may also aggravate the existing systemic disease by changing the inflammatory parameters in the body. The aim of this study was to evaluate the effect of obesity and exercise on periodontal and biochemical parameters [serum, saliva and gingival crevicular fluid (GCF) adipokines (interleukin-1β, tumor necrosis factor-α, leptin, resistin and adiponectin)].

ELIGIBILITY:
Inclusion Criteria:

* Being women,
* Older than 18 yrs old,
* Not being pregnant,
* Not being disabled,
* For study group; being obese, not for healthy group being systemically health and in normal weight
* Not treated periodontological in the last 6 months

Exclusion Criteria:

* Younger than 18 yrs old,
* Smokers who smokes more than 10 cigarettes in a day,
* Uncontrolled systemic diseases,
* Having periodontal treatment
* who needs antibiotic prophylaxis

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — adult women
Enrollment: 71 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2016-01-10 (Actual)

PRIMARY OUTCOMES:
Biochemical variables GCF | 12 week
  TNF-A, IL-1B,concentrations levels (pg/µl)
Biochemical variables GCF | 12 week
  Leptin, adiponectin, resistin concentrations levels (ng/µl)

SECONDARY OUTCOMES:
Biochemical variables_Saliva | 12 week
  TNF-A, IL-1B,concentrations levels (pg/µl)
Biochemical variables_Saliva | 12 week
  leptin, adiponectin, resistin concentrations levels (ng/µl)
Biochemical variables_Serum | 12 week
  TNF-A, IL-1B,concentrations levels (pg/µl)
Biochemical variables_Serum | 12 week
  leptin, adiponectin, resistin concentrations levels (ng/µl)

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided